CLINICAL TRIAL: NCT02249247
Title: Effect of 12-week Treatment of 5, 25 or 75 mg BIIL 284 BS on Exercise Endurance in Patients With Chronic Obstructive Pulmonary Disease (Double-blind, Double Dummy, Placebo-controlled, Randomized, Parallel Group, Dose Ranging Study)
Brief Title: Effect of Treatment With BIIL 284 BS on Exercise Endurance in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.17
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — amelubant

ARMS (4):
- Low dose of BIIL 284 BS (Experimental)
  Interventions: Drug: Low dose of BIIL 284 BS tablets
- Medium dose of BIIL 284 BS (Experimental)
  Interventions: Drug: Medium dose of BIIL 284 BS tablets
- High dose of BIIL 284 BS (Experimental)
  Interventions: Drug: High dose of BIIL 284 BS tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of BIIL 284 BS tablets
  Arms: Low dose of BIIL 284 BS
Drug: Medium dose of BIIL 284 BS tablets
  Arms: Medium dose of BIIL 284 BS
Drug: High dose of BIIL 284 BS tablets
  Arms: High dose of BIIL 284 BS
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate the effect of 12-week treatment with three doses (5, 25 and 75 mg) BIIL 284 BS on exercise endurance, lung function, quality of life, spontaneous sputum and safety in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD as defined by the American Thoracic Society (ATS) criteria. Patients had to have relatively stable airway obstruction with a FEV1 ≥ 20 % and ≤ 70 % of predicted value and FEV1/ FVC ≤ 70 % at screening Visit 1. Predicted normal values were based on the guidelines for standardised lung function testing of the European Community for Steel and Coal (ECSC) for patients of the Caucasian race and on the predicted equations for patients belonging to the Black race. Patients had to have lung hyperinflation as demonstrated by thoracic gas volume box (TGVbox) ≥ 100 % of predicted value (same as predicted value for functional residual capacity (FRC) measured by body plethysmography)
* Males or females aged 40 years or older. Female patients of childbearing potential could not participate in this study. Female patients had to be either:

  * surgically sterilised by hysterectomy or bilateral tubal ligation, or
  * post-menopausal for at least two years
* A smoking history of more than ten pack-years (p.y.). A p.y. was defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
* Patients had to be able to perform pulmonary function testings (PFTs), exercise endurance test not terminated due to leg discomfort alone or other restrictions diseases (e.g. claudicatio intermittens, etc.) only and maintain records during the study period as required in the protocol
* All patients had to sign both informed consent forms (one on specific study procedures, one related to DNA derived determinations) prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications if they agreed to participate in both portions of the trial. The patient was not obligated to participate in the DNA collection portion of the trial

Exclusion Criteria:

* Clinical and/or radiographic evidence and/or antibiotic treatment of an upper or lower respiratory tract infection within the previous four weeks or during the screening period of this study
* Significant diseases other than COPD were excluded. A significant disease was defined as a disease which in the opinion of the investigator could either put the patient at risk because of participation in the study or a disease which could influence the results of the study or the patient's ability to participate in the study. Patients with inflammatory diseases, e.g., Rheumatoid Arthritis (RA), osteoarthritis, and those with autoimmune diseases were excluded
* Clinically significant abnormal baseline haematology, liver function, blood chemistry or urinalysis. If the abnormality defined a disease listed as an exclusion criterion the patient was excluded
* A recent history (i.e., within six months) of myocardial infarction
* A recent history (i.e., within three months) of refractory heart failure or unstable arrhythmia requiring treatment
* Patients with known tuberculosis
* A history of cancer within the last five years. Patients with treated basal cell carcinoma or cutaneous squamous cell carcinoma were allowed
* A history of life-threatening airway obstruction or a history of cystic fibrosis
* Previous thoracotomy with pulmonary resection. Patients with a history of a thoracotomy without pulmonary resection were evaluated as per exclusion criterion No. 2
* A change in pulmonary therapy, including rehabilitation therapy, within the four weeks prior to the first screening Visit (Visit 1) in order to control the patient's COPD
* A history of asthma or a total blood eosinophil count ≥ 600/mm3. A repeat eosinophil count was not conducted in these patients
* A history (within the past five years) of and/or current alcohol abuse and/or drug abuse
* Use of an investigational drug within one month or six half lives (which ever is greater) of the first Screening Visit (Visit 1)
* Patients requiring oxygen therapy 24 hours a day or requiring oxygen during exercise. Patients that desaturated during exercise were only excluded upon medical judgement of the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2001-04; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Changes in exercise endurance | Pre-dose, up to 12 weeks after start of treatment
  evaluated by constant work load test

SECONDARY OUTCOMES:
Changes in breathlessness during constant work load test | Week 4 and week 12 weeks after start of treatment
  measured by Modified Borg scale: Dyspnea score, leg discomfort
Changes in forced expiratory volume in one second (FEV1) | Pre-dose, up to 12 weeks after start of treatment
  assessed by spirometry
Changes in forced vital capacity (FVC) | Pre-dose, up to 12 weeks after start of treatment
  assessed by spirometry
Changes in forced expiratory flow at 25%-75% of FVC (FEF25-75%) | Pre-dose, up to 12 weeks after start of treatment
  assessed by spirometry
Changes in inspiratory capacity (IC) | Pre-dose, up to 12 weeks after start of treatment
  assessed by spirometry
Changes in slow vital capacity (SVC) | Pre-dose, up to 12 weeks after start of treatment
  assessed by spirometry
Change in thoracic gas volume | Pre-dose, up to 12 weeks after start of treatment
  assessed by body plethysmography
Changes in total lung capacity | Pre-dose, up to 12 weeks after start of treatment
  assessed by body plethysmography
Changes in residual volume | Pre-dose, up to 12 weeks after start of treatment
  assessed by body plethysmography
Changes in specific airway conductance | Pre-dose, up to 12 weeks after start of treatment
  assessed by body plethysmography
Changes in Mahler dyspnoea questionnaire | Pre-dose, up to 12 weeks after start of treatment
  Baseline dyspnoea index / transitional dyspnoea index (BDI/TDI)
Changes in chronic respiratory disease questionnaire (CRDQ) | Pre-dose, up to 12 weeks after start of treatment
Changes in carbon monoxide diffusing capacity (DLco) | Pre-dose, up to 12 weeks after start of treatment
Changes in diffusing capacity of carbon monoxide corrected for alveolar volume (DLco/VA) | Pre-dose, up to 12 weeks after start of treatment
Changes in peak expiratory flow rate (PEFR) daily patient record | Pre-dose, up to 14 weeks after start of treatment
  assessed a.m. and p.m. in daily patient record
Changes in 24-hours spontaneous sputum wet weight | Pre-dose, up 12 weeks after start of treatment
Changes in oxygen saturation during constant work load test | Pre-dose, up to 12 weeks after start of treatment
  assessed by pulse oximetry
Changes in global evaluation assessed by investigator on a 4-point scale | Pre-dose, up to 14 weeks after start of treatment
Clinically relevant changes in vital signs (pulse rate, blood pressure) | Pre-dose, up to 14 weeks after start of treatment
Clinically relevant changes in ECG | Pre-dose, up to 14 weeks after start of treatment
Clinically relevant changes in laboratory tests | Pre-dose, up to 14 weeks after start of treatment
Number of patients with adverse events | Up to 17 weeks
Number of patients with acute COPD exacerbations | Up to 17 weeks